CLINICAL TRIAL: NCT04318314
Title: COVID-19: Healthcare Worker Bioresource: Immune Protection and Pathogenesis in SARS-CoV-2
Acronym: COVID19-HCW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: St. Bartholomew's Hospital (Other); Royal Free Hospital NHS Foundation Trust (Other); UCLH (Unknown)
Responsible Party: Sponsor
Other Study IDs: 130852
Record Dates: First submitted 2020-03-17; First posted 2020-03-23 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Health Care Worker Patient Transmission; Coronavirus; Coronavirus Infections; Immunological Abnormality
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood samples Nasal and oropharygeal swabs Saliva samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy and asymptomatic healthcare workers: Healthy and asymptomatic healthcare workers
  Interventions: Diagnostic Test: COPAN swabbing and blood sample collection

INTERVENTIONS:
Diagnostic Test: COPAN swabbing and blood sample collection — COPAN swabbing of nostrils and/or oropharynx and blood sample collection

SUMMARY:
Modelling repurposed from pandemic influenza is currently informing all strategies for SARS-CoV-2 and the disease COVID-19. A customized disease specific understanding will be important to understand subsequent disease waves, vaccine development and therapeutics. For this reason, ISARIC (the International Severe Acute Respiratory and Emerging Infection Consortium) was set up in advance. This focuses on hospitalised and convalescent serum samples to understand severe illness and associated immune response. However, many subjects are seroconverting with mild or even subclinical disease. Information is needed about subclinical infection, the significance of baseline immune status and the earliest immune changes that may occur in mild disease to compare with those of SARS-CoV-2. There is also a need to understand the vulnerability and response to COVID-19 of the NHS workforce of healthcare workers (HCWs). HCW present a cohort with likely higher exposure and seroconversion rates than the general population, but who can be followed up with potential for serial testing enabling an insight into early disease and markers of risk for disease severity. We have set up "COVID-19: Healthcare worker Bioresource: Immune Protection and Pathogenesis in SARS-CoV-2". This urgent fieldwork aims to secure significant (n=400) sampling of healthcare workers (demographics, swabs, blood sampling) at baseline, and weekly whilst they are well and attending work, with acute sampling (if hospitalised, via ISARIC, if their admission hospital is part of the ISARIC network) and convalescent samples post illness. These will be used to address specific questions around the impact of baseline immune function, the earliest immune responses to infection, and the biology of those who get non-hospitalized disease for local research and as a national resource. The proposal links directly with other ongoing ISARIC and community COVID projects sampling in children and the older age population. Reasonable estimates suggest the usable window for baseline sampling of NHS HCW is closing fast (e.g. baseline sampling within 3 weeks).

DETAILED DESCRIPTION:
The proposed study is a prospective observational cohort design which will be carried out across three different trusts: Barts Health NHS Trust (St Bartholomew's Hospital, The Royal London Hospital, Whipps Cross Hospital and Newham Hospital), Royal Free London NHS Foundation Trust (Royal Free Hospital) and University College London Hospitals NHS Foundation Trust (UCLH).

Participants will be asymptomatic front-facing HCWs who carry out their tasks in different areas of the corresponding hospital: Accident and Emergency, Adult Medical Admissions Unit, Medical and Surgical Wards and Intensive Care Units.

This study substantially uses existing infrastructure: Recruits into this study who are subsequently suspected to have COVID-19 can be co-recruited into ISARIC using ISARIC Ethics Ref: 13/SC/0149 (Oxford C Research Ethics Committee, UK CRN /CPMS ID 14152 IRAS ID126600 for acute samples and data collection. Sampling can be delivered via existing research personnel from furloughed projects (CLRN nurses, research fellows, Barts Bioresource). Convalescent sampling will be via an otherwise inactive Clinical Trials unit. It

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years AND
* Asymptomatic (meaning healthy enough to attend work according to Trust policy at the time) AND
* Work in the designated clinical environments for at least 5 hours for at least one day during the study period.

Participants will be free to withdraw from the study at any point, but collection of these data is considered to be in the public interest and will fall under the scope of a 'Public task' by the GDPR definition. Under these conditions rights to erasure and data portability do not apply, and archiving and further processing for scientific research purposes is compatible with the original purpose; no further participant data from medical records will be collected.

The research team may withdraw a participant from the study in the following situations:

- No longer meets the inclusion/exclusion criteria if participants circumstance change

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy asymptomatic healthcare workers attending their usual place of work that can be St Bartholomew's Hospital, Royal Free London or UCLH.
Sampling Method: Non-Probability Sample
Enrollment: 731 (Estimated)
Dates: Start 2020-03-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion to SARS-CoV-2 positivity | Within 12 months
  Home-isolation or hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: James C Moon, Principal Investigator — BHC & UCL; Charlotte Manisty, Study Director — BHC & UCL; Thomas Treibel, Principal Investigator — Barts Heart Center
Locations (2):
- United Kingdom (2):
  - Barts Heart Center, London
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Publication of results in open access journals; sharing of results in scientific databases.
Supporting Information: Study Protocol, ICF
Time Frame: 24 months
URL: https://covid-consortium.com

REFERENCES:
- [Derived] Altmann DM, Reynolds CJ, Joy G, Otter AD, Gibbons JM, Pade C, Swadling L, Maini MK, Brooks T, Semper A, McKnight A, Noursadeghi M, Manisty C, Treibel TA, Moon JC; COVIDsortium investigators; Boyton RJ. Persistent symptoms after COVID-19 are not associated with differential SARS-CoV-2 antibody or T cell immunity. Nat Commun. 2023 Aug 23;14(1):5139. doi: 10.1038/s41467-023-40460-1. PMID 37612310
- [Derived] Wing PAC, Schmidt NM, Peters R, Erdmann M, Brown R, Wang H, Swadling L; COVIDsortium Investigators; Newman J, Thakur N, Shionoya K, Morgan SB, Hinks TS, Watashi K, Bailey D, Hansen SB, Davidson AD, Maini MK, McKeating JA. An ACAT inhibitor suppresses SARS-CoV-2 replication and boosts antiviral T cell activity. PLoS Pathog. 2023 May 3;19(5):e1011323. doi: 10.1371/journal.ppat.1011323. eCollection 2023 May. PMID 37134108
- [Derived] Doykov I, Baldwin T, Spiewak J, Gilmour KC, Gibbons JM, Pade C, Reynolds CJ, Aine McKnight, Noursadeghi M, Maini MK, Manisty C, Treibel T, Captur G, Fontana M, Boyton RJ, Altmann DM, Brooks T, Semper A; UK COVIDsortium Investigators; Moon JC, Kevin Mills, Heywood WE. Quantitative, multiplexed, targeted proteomics for ascertaining variant specific SARS-CoV-2 antibody response. Cell Rep Methods. 2022 Sep 19;2(9):100279. doi: 10.1016/j.crmeth.2022.100279. Epub 2022 Aug 12. PMID 35975199
- [Derived] Astbury S, Reynolds CJ, Butler DK, Munoz-Sandoval DC, Lin KM, Pieper FP, Otter A, Kouraki A, Cusin L, Nightingale J, Vijay A, Craxford S, Aithal GP, Tighe PJ, Gibbons JM, Pade C, Joy G, Maini M, Chain B, Semper A, Brooks T, Ollivere BJ, McKnight A, Noursadeghi M, Treibel TA, Manisty C, Moon JC; COVIDsortium Investigators*; Valdes AM, Boyton RJ, Altmann DM. HLA-DR polymorphism in SARS-CoV-2 infection and susceptibility to symptomatic COVID-19. Immunology. 2022 May;166(1):68-77. doi: 10.1111/imm.13450. Epub 2022 Mar 8. PMID 35156709
- [Derived] Valdes AM, Moon JC, Vijay A, Chaturvedi N, Norrish A, Ikram A, Craxford S, Cusin LML, Nightingale J, Semper A, Brooks T, McKnight A, Kurdi H, Menni C, Tighe P, Noursadeghi M, Aithal G, Treibel TA, Ollivere BJ, Manisty C. Longitudinal assessment of symptoms and risk of SARS-CoV-2 infection in healthcare workers across 5 hospitals to understand ethnic differences in infection risk. EClinicalMedicine. 2021 Apr;34:100835. doi: 10.1016/j.eclinm.2021.100835. Epub 2021 Apr 15. PMID 33880438

DOCUMENTS (3):
  • Study Protocol: List of Publications (2021-05-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT04318314/Prot_000.pdf
  • Study Protocol: Last Amendment N 4 - Description and Approval Letter (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT04318314/Prot_001.pdf
  • Study Protocol: Full Study Protocol Updated 21/09/2020 (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT04318314/Prot_002.pdf